CLINICAL TRIAL: NCT04175756
Title: CAIman 5 Articulating Maryland in coloRECTAL Cancer Surgery. An Observational, Prospective, Post-marketing Clinical Follow-up Study
Brief Title: CAIman 5 Articulating Maryland in coloRECTAL Cancer Surgery
Acronym: CAIRECTAL
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1627
Record Dates: First submitted 2019-11-19; First posted 2019-11-25 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; laparoscopic surgery; Seal & Cut; Total Mesorectal Excision (TME); Partial Mesorectal Excision (PME); Complete Mesocolic Excision (CME)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Caiman 5 articulating Maryland — Laparoscopic colorectal surgery

SUMMARY:
This voluntary study is part of a Post-Market-Surveillance plan to proactively collect clinical data for the use of Caiman 5 articulating Maryland in colorectal surgery under daily clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Patient´s written informed consent
* Planned laparoscopic colorectal cancer surgery using Caiman 5 articulating Maryland (according to the IfU)
* Age ≥18 years

Exclusion Criteria:

* Emergency surgery
* Pregnancy
* Participation in another surgical study, which might influence the intraoperative process
* Conversion to open surgery
* Conversion to another sealing / cutting instrument (instead of Caiman 5 articulating Maryland)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Total operative time | intraoperatively
  Time between first incision and closure of the surgical incision

SECONDARY OUTCOMES:
Complications | up to 4 months postoperative
  Number of Complications: Wound infections, Urinary tract infections, Pulmonary infections, Other infections, Wound dehiscence, Anastomotic leak, Anastomotic bleeding, Other bleeding / hemorrhage, Intraabdominal abscess, Fistula, Peritonitis, Sepsis, Hernia, Stenosis Ileus, Ureter injury, Nerve injury, Cardiac complications, Other
Handling characteristics | intraoperative
  Evaluation of performance and handling characteristics using a questionnaire containing 5-level Likert scales (excellent, very good, good, fair, poor)
Estimated intraoperative blood loss | intraoperative
  intraoperative blood loss in ml
Time needed for TME | Intraoperative
  Time between end of left flexure mobilization and stapling
Time needed for PME | Intraoperative
  Time [in minutes] between end of left flexure mobilization and stapling
Time needed for CME | Intraoperative
  Time [in minutes] between end of ileocolic vessels clipping and start of right flexure mobilization
Time needed for right / hepatic colic flexure mobilization | Intraoperative
  Time [in minutes] between end CME and start of resection of the mesentery of the small intestine
Time needed for left / splenic colic flexure mobilization | Intraoperative
  Time [in minutes] between clipping of inferior mesenteric vessels and start of TME, PME or corresponding)
Stay in intensive care unit postop | up to discharge (approximately 10 days postoperative)
  Number of days postoperative until discharge from intensive care unit
Stay in intermediate care unit stay postop | up to discharge (approximately 10 days postoperative)
  Number of days postoperative until discharge from intermediate care unit stay
First postoperative oral intake | up to discharge (approximately 10 days postoperative)
  Number of days until patient's first postoperative oral intake
First postoperative stool | up to discharge (approximately 10 days postoperative)
  Number of days until patient's first postoperative stool after oral intake
Quality of excision: M.E.R.C.U.R.Y. criteria | up to discharge (approximately 10 days postoperative)
  quality of mesorectal excision according to criteria established in the "Magnetic Resonance Imaging and Rectal Cancer European Equivalence Study" (M.E.R.C.U.R.Y.)

CONTACTS AND LOCATIONS:
Overall Officials: Niedergethmann, Prof. Dr. med., Principal Investigator — Alfried Krupp Krankenhaus, 45131 Essen
Locations (1):
- Alfried Krupp Krankenhaus Rüttenscheid, Essen, Germany